CLINICAL TRIAL: NCT05518591
Title: A Randomised Control Trial Comparing Compassion Focused Therapy and Breathing Pattern Retraining With Treatment as Usual in Patients Diagnosed With Cancer Recurrence During COVID.
Brief Title: COMpassion FOcused Therapy and Breathing Pattern REtraining After Cancer Recurrence
Acronym: COMFORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other); Irish Cancer Society (Other)
Responsible Party: Principal Investigator, Donal Brennan, Professor Donal Brennan, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COV21LYN
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Psychological Distress; Cancer Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CFT & BPR (Experimental): 6-week, virtual, psychological therapy group involving compassion focused therapy and breathing pattern retraining. This group involves exercises in practicing self-compassion, emotional regulation, and breathing retraining.
  Interventions: Behavioral: Compassion Focused Therapy (CFT) combined with Breathing Pattern Retraining (BPR)
- Treatment As Usual (No Intervention): Those in the treatment as usual arm are not being asked to engage in anything additional to their regular treatment plan. They will, however, be given the option to participate in the psychological intervention after the study has ended, if they elect to do so.

INTERVENTIONS:
Behavioral: Compassion Focused Therapy (CFT) combined with Breathing Pattern Retraining (BPR) — Study participants in the experimental arm of the study are being asked to take part in a 6-week, virtual, psychological therapy group involving compassion focused therapy and breathing pattern retraining. This group involves exercises in practicing self-compassion, emotional regulation, and breathing retraining. Each group session lasts less than two hours, per week.
  Arms: CFT & BPR

SUMMARY:
The purpose of this study is to investigate how effective a particular psychological intervention is at reducing psychological distress for people who were diagnosed with cancer 'recurrence' since the beginning of the COVID pandemic.

DETAILED DESCRIPTION:
This study plans to study how effective a particular psychological intervention is at reducing psychological distress for people who were diagnosed with cancer 'recurrence' since the beginning of the pandemic, having previously been diagnosed with cancer. We know that a cancer diagnosis can often result in significant psychological distress. After or during treatment for cancer, individuals often experience a 'fear of recurrence', which should it occur, often results in a state of mental anguish that is described as being more punishing than the initial diagnosis itself. Being diagnosed with a cancer recurrence diagnosis can trigger marked negative psychological symptoms, including distress, uncertainty, traumatic distress and adjustment problems, with psychological recovery from this diagnosis often being slower than that of the initial cancer diagnosis. The COVID-19 pandemic has affected these patients further, in terms of restricted access to healthcare, reduced social supports, and greater levels of treatment uncertainty. Our research team has designed a psychological intervention that is specifically aimed to help some of these issues. It's a 6-week online group intervention using a 'compassion focused therapy' approach, coupled with specialised breathing techniques to reduce bodily distress. It is being done online due to ongoing concerns around COVID but also to eliminate geographical and/or commuting barriers. It is our expectation that those receiving the psychological intervention will experience noticeable reductions in measures of psychological distress compared to those who are receiving regular treatment. It is our hope that the outcomes of this study will inform how best to help patients facing into cancer recurrence at a national level.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 or older
* pre-existing cancer diagnosis
* diagnosis of cancer recurrence during COVID-19 (March 2020 onwards)
* Living in Ireland
* English speaking / fluency
* Access to web / tech support

Exclusion Criteria:

* A score <4 on the Distress Thermometer
* Patient non-consent
* The presence of a severe mental illness (such as schizophrenia, personality disorder or active illness)
* Known or suspected drug or alcohol abuse problems within past 3 months
* Inability to follow the study procedures e.g. dementia or non-fluency of English
* Life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Overall Distress Score | 12 weeks post completion of intervention
  The primary outcome is the patient's overall distress score, based on the Distress Thermometer (DT)

SECONDARY OUTCOMES:
Changes in depressive symptoms | 12 weeks post completion of intervention
  Patient Health Questionnaire-9 (PHQ-9) will assesses symptoms of depression
Changes in anxiety symptoms | 12 weeks post completion of intervention
  General Anxiety Disorder-7 (GAD-7) will assesses symptoms of anxiety
Changes in traumatic distress | 12 weeks post completion of intervention
  Impact of Event Scales- Revised (IES-R) will measure the amount of distress that a subject associates with a specific event.
Mental Adjustment to Cancer Recurrence | 12 weeks post completion of intervention
  Mini-Mental Adjustment to Cancer (MAC) scale will measure a subjects ability to cope with diagnosis of recurrence and and assesses five cancer-specific coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Lynch, PhD, Principal Investigator — MMUH
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynch S, Lowry D, Finnerty C, O'Meara Y, Brennan D. The COMFORT trial: a randomised control trial comparing group-based COMpassion-FOcussed therapy and breathing pattern ReTraining with treatment as usual on the psychological functioning of patients diagnosed with cancer recurrence during COVID. Trials. 2023 Feb 6;24(1):89. doi: 10.1186/s13063-023-07088-4. PMID 36747246